CLINICAL TRIAL: NCT06145633
Title: Vorinostat to Augment Response to 177Lutetium-PSMA-617 in the Treatment of Patients With PSMA-Low Metastatic Castration-Resistant Prostate Cancer
Brief Title: Vorinostat and 177Lu-PSMA-617 for the Treatment of PSMA-Low Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Novartis (Industry); Institute for Prostate Cancer Research (IPCR) (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123920; NCI-2023-08921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020244 (Other: Fred Hutch/University of Washington Cancer Consortium); R37CA286450 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Fluorodeoxyglucose F18; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Pluvicto; Magnetic Resonance Spectroscopy; X-Rays; Photons; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vorinostat, 177Lu-PSMA-617) (Experimental): Patients receive vorinostat PO QD for 28 days and then receive gallium Ga 68 gozetotide IV and undergo a PET scan on trial. Patients may go on to receive 177Lu-PSMA-617 IV per SOC on day 1 of each cycle. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT and bone scan on trial and during follow-up, as well as a FDG PET/CT during screening and on trial and SPECT/CT on trial. Patients undergo blood sample collection on trial and may also optionally undergo biopsy during screening and on trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography; Drug: Vorinostat

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT, PET/CT, SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given 177Lu-PSMA-617
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Positron Emission Tomography — Undergo 68Ga-PSMA-11 PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Drug: Vorinostat — Given IV
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial tests how well vorinostat works in treating patients with prostate-specific membrane antigen (PSMA)-low castration-resistant prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic) (mCRPC). Prostate cancer that has not spread to other parts of the body (localized) is typically treated through surgery or radiotherapy, which for many men is curable. Despite definitive local therapy, cancer that has come back after a period of improvement (recurrent) disease develops in 27-53% of men. Often this is detected by measurement of prostate-specific antigen (PSA) without visible evidence of metastatic disease. Lutetium Lu 177 vipivotide tetraxetan (177Lu-prostate specific membrane antigen [PSMA]-617) is a new small molecule PSMA-targeted radioactive therapy that has been approved by the Food and Drug Administration for the treatment of adult patients with PSMA-positive mCRPC who have been treated with androgen receptor inhibitors and taxane-based chemotherapy. Vorinostat is used to treat various types of cancer that does not get better, gets worse, or comes back during or after treatment with other drugs. Vorinostat is a drug which inhibits the enzyme histone deacetylase and may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat and 177Lu-PSMA-617 may kill more tumor cells in in patients with PSMA-low mCRPC.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive vorinostat orally (PO) once a day (QD) for 28 days and then receive gallium Ga 68 gozetotide intravenously (IV) and undergo a positron emission tomography (PET) scan on trial. Patients may go on to receive 177Lu-PSMA-617 IV per standard of care (SOC) on day 1 of each cycle. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) and bone scan on trial and during follow-up, as well as a fludeoxyglucose F-18 (FDG) PET/CT during screening and on trial and single photon emission computed tomography (SPECT)/CT on trial. Patients undergo blood sample collection on trial and may also optionally undergo biopsy during screening and on trial.

After completion of study treatment, patients are followed up every 8 weeks for 6 months and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically confirmed adenocarcinoma of the prostate.
* Patient must have evidence of castration resistant prostate cancer as evidenced by PSA progression (per Prostate Cancer Working Group 3 [PCWG3] criteria) and a castrate serum testosterone level (i.e., ≤ 50 mg/dL).
* PSMA SUVmean < 10 as determined by 68Ga-PSMA-11 PET.
* Patients must have received a next-generation androgen receptor-signaling inhibitor (e.g. abiraterone, enzalutamide, apalutamide, darolutamide). There must be at least a 2-week washout period after stopping these agents. Patients should be weaned off steroids at least 1 week prior to starting treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT and/or bone scan and is suitable for repeated assessment.
* Hemoglobin ≥ 10 g/dL (measured within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Platelet count ≥ 100 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN (measured within 28 days prior to administration of study treatment) . For patients with known Gilbert's Syndrome they must be ≤ 3 x ULN (measured within 28 days prior to administration of study treatment)
* Calculated creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula) (measured within 28 days prior to administration of study treatment)
* Patients and their partners, who are sexually active and of childbearing potential must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 3 months after last dose of study drug to prevent pregnancy in a partner.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition that could interfere with patient safety or provision of informed consent to participate in this study.
* Evidence of metastatic neuroendocrine/small cell prostate cancer (NEPC). Note: baseline biopsy is not required but is strongly encouraged if a patient is found to have an FDG-positive/PSMA-negative lesion on baseline imaging.
* Patients receiving any systemic therapy (aside from an luteinizing hormone-releasing hormone [LHRH] analogue) or radiotherapy within 2 weeks prior to study treatment.
* Any previous treatment with an HDAC inhibitor (including valproic acid) or 177Lu-PSMA-617.
* Persistent toxicities (CTCAE grade >2) from prior cancer therapy, excluding alopecia and stable neuropathy.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder or active, uncontrolled infection. Examples include, but are not limited to uncontrolled seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Patients who are known to be serologically positive for human immunodeficiency virus (HIV) and a CD4 count < 200.
* Patients with known active hepatitis (i.e. Hepatitis B or C). Prior Hep C infection is allowed as long as polymerase chain reaction (PCR) is negative.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Deep vein thrombosis or pulmonary embolism diagnosed within the past six months.
* Active use of coumarin-derived anticoagulant medication (i.e. warfarin).
* Serious cardiac disorder, including but not limited to uncontrolled ventricular arrhythmia, recent (within 12 months) myocardial infarction, resting electrocardiogram (ECG) indicating Fridericia's corrected QT interval prolongation > 500ms, or congenital long QT syndrome.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who convert from prostate-specific membrane antigen (PSMA) low to PSMA high | Up to 40 weeks
  Will be calculated as the percentage with 95% confidence interval (CI) of the total number of patients who had PSMA-high expression on re-assessment gallium Ga 68 gozetotide (68Ga)-PSMA-11 positron emission tomography (PET).

SECONDARY OUTCOMES:
Objective radiographic response rate | Up to 2 years
  Will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Prostate specific antigen (PSA)50 response rate | Baseline up to 2 years
  The percent decline in PSA compared to baseline (the PSA level prior to initiation of lutetium Lu 177 vipivotide tetraxetan will be calculated for each patient for every on-study PSA value obtained. PSA50 response will be defined as a decline in PSA ≥ 50% compared to baseline. Will be reported as a percentage with 95% CI.
Progression free survival (PFS) | From the start of treatment until disease progression, clinical progression, or death, whichever occurs first, assessed up to 2 years
  Disease progression measured by modified RECIST criteria or Prostate Cancer Working Group 3 criteria for bone lesions and clinical progression as determined by the treating physician. Will be estimated using Kaplan-Meier method.
PSA PFS | From the start of treatment until PSA progression, assessed up to 2 years
  For patients showing an initial decline in PSA from baseline, PSA progression will be defined as an increase in PSA ≥ 25% and ≥ 2 ng/mL above the nadir, and which is confirmed by a second value 3 or more weeks later. For those with no decline in PSA from baseline, PSA progression will be defined as an increase in PSA that is ≥ 25% and ≥ 2ng/mL after 12 weeks. Will be estimated using Kaplan-Meier method.
Overall survival | From the start of treatment until death from any cause, assessed up to 2 years
  Will be estimated using Kaplan-Meier method.
Number of discrete lesions | Up to 40 weeks
  Will determine the number of discrete lesions on imaging converted from low to high PSMA expression across the study population at the time of re-assessment 68Ga-PSMA-11 PET.
Absolute change in PSMA standardized uptake value (SUV) mean | Up to 40 weeks
  PSMA SUVmean will be determined by an experienced nuclear medicine physician by measuring the PSMA SUV at each site of PSMA positive disease and dividing by the total PSMA positive tumor volume.
Incidence of adverse events | Up to 2 years
  Will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Event version 5.0 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No